CLINICAL TRIAL: NCT05051995
Title: Combined N-of-1 Trials to Assess Open-Label Placebo Treatment for Antidepressant Discontinuation Symptoms
Acronym: FAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Philipps University Marburg (Other); Helmut Schmidt University (Other); University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0721-20; CRC 289 Project A15 (Other Grant/Funding Number: DFG Deutsche Forschungsgemeinschaft); U1111-1274-2336 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2021-08-23; First posted 2021-09-21 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Depressive Symptoms; Expectations; Antidepressants
Keywords: N-of-1 trials; open-label placebo; discontinuation symptoms; antidepressant medication; expectation effects
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: To investigate the efficacy of open-label placebo in the reduction of antidepressant discontinuation symptoms, patients experiencing moderate discontinuation symptoms after successful discontinuation (4 weeks) receive open-label placebo treatment or no treatment during the experimental phase (8 weeks).
  For this purpose, a series of N-of-1 trials is implemented, consisting of multiple crossover trials within each participant. The factor treatment (open-label placebo vs. no treatment) varies intra-individually with a biweekly rhythm, to assess the treatment effect on discontinuation symptoms. A block-randomization is applied, with patients either receiving (A) open-label placebo or (B) no treatment in a biweekly rhythm (group 1: ABAB; group 2: BABA).
Who Masked: Outcomes Assessor
Masking Description: The person performing the data collection (assessor) will be blind to the randomization of the participant for the entire duration of the experimental phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-label placebo ABAB Sequence (Placebo Comparator): The N-of-1 trial will, on the level of the individual patient, test whether open-label placebo reduces negative side effects caused by discontinuation of antidepressants compared to no treatment. After antidepressant discontinuation, subjects will be randomized to 2 arms differing in the treatment order (ABAB; BABA). Subjects in this arm (ABAB) will start with open-label placebo (A) for 2 weeks; they will then crossover to no treatment (B) for 2 weeks and repeat this sequence once again.
  Interventions: Drug: Open-label placebo; Other: No-treatment
- Open-label placebo BABA Sequence (Placebo Comparator): The N-of-1 trial will, on the level of the individual patient, test whether open-label placebo reduces negative side effects caused by discontinuation of antidepressants compared to no treatment. After antidepressant discontinuation, subjects will be randomized to 2 arms differing in the treatment order (ABAB; BABA). Subjects in this arm (BABA) will start with no treatment (B) for 2 weeks; they will then crossover to open-label placebo (A) for 2 weeks and repeat this sequence once again.
  Interventions: Drug: Open-label placebo; Other: No-treatment

INTERVENTIONS:
Drug: Open-label placebo — Prior to the open-label placebo administration, an explanation why placebos without concealment might be effective is offered. Participants receive placebo pills with the instruction to take 2 pills daily for 2 weeks.
Other: No-treatment — During the no-treatment phase, participants receive no treatment for 2 weeks.

SUMMARY:
It has been widely recognized that the placebo effect has a profound impact on treatment outcome in many different conditions. Recent studies imply that this effect appears even if placebos are openly administered; so called "open-label placebos" (OLP). Compelling evidence suggests the efficacy of OLP in the treatment of pain disorders, neuropsychological syndromes, menopausal hot flushes, depression and allergic rhinitis. Research on the underlying mechanisms of OLP is scarce, yet studies indicate that psychological mechanisms as well as neurobiological processes related to expectation- and prediction mechanisms may play a role. While these effects have been linked to OLP as additional treatment, to date, it has not been examined whether OLP could support discontinuation of drug treatments.

Antidepressant discontinuation has been frequently associated with negative side effects, interfering with the discontinuation process and generally discouraging discontinuation. Patients frequently report negative expectations towards the discontinuation process, such as fear of experiencing a relapse and negative side effects. Interestingly, OLP may support antidepressant discontinuation, not only through the generation of (positive) expectations, but also mechanisms related to habituation (i.e. taking pills). The objective of this study is to investigate whether OLP is efficacious in reducing negative side effects caused by discontinuation of antidepressant medication.

This preregistration is part of the collaborative research center (CRC) SFB/ TRR289 which aims to characterize the psychological and neurobiological effects of treatment expectations on health outcome (https://treatment-expectation.de) and is funded by the Deutsche Forschungsgemeinschaft (DFG).

DETAILED DESCRIPTION:
Rationale: A current issue in the frame of antidepressant medication is the rise of long-term antidepressant use associated with noticeable adverse effects such as withdrawal effects, sexual difficulties, weight gain and emotional numbness. A key factor hindering patients in the discontinuation of antidepressant medication is the emergence of discontinuation symptoms, reported by over half of fully remitted patients discontinuing antidepressants. To date, there is no study examining open-label placebo responses on antidepressant discontinuation symptoms. However, several findings imply that open-label placebos may support the discontinuation process in remitted depressed patients. The susceptibility to placebo responses is encouraged by findings indicating substantial placebo effects in antidepressant trials (67-82%). Additionally, evidence suggests the central role of expectation effects influencing the course of antidepressant discontinuation. Open-label placebos have been found to work through the generation of positive expectations, induced by a positive framing (e.g. verbal instructions). A recent meta-analysis suggests a medium to large effect size of open-label placebos. Regarding the treatment of antidepressant discontinuation symptoms, open-label placebos have the potential to reduce symptoms not only by inducing positive expectations, but also by triggering automatic (positive) responses to the intake of a pill (i.e. conditioning).The aim of this study is to investigate the effect of open-label placebos on antidepressant discontinuation symptoms in fully remitted depressed patients.

Methods: In the proposed study, a pilot sample will discontinue their antidepressant intake under extensive medical and psychological supervision, according to the national and international guidelines over a 13-week course. After a run-in week and the baseline assessment, antidepressant medication will be gradually reduced with individualized discontinuation plans over a period of 4 weeks. Weekly measurements serve to monitor the condition of the participants. After discontinuation, patients will be monitored (with biweekly study visits) for another 8 weeks (experimental phase). Finally, a follow-up measurement 6 months after the study start constitutes long-term monitoring and the assessment of relapse after antidepressant discontinuation. During the experimental phase, patients experiencing moderate discontinuation symptoms are allocated to the intervention group, aimed to examine the effect of open-label placebo on antidepressant discontinuation symptoms. For this purpose, N-of-1 trials comprising multiple crossovers (A: open-label placebo; B: no treatment) within each individual, and varying in a biweekly rhythm, are applied. Patients are randomized to different treatment orders (ABAB; BABA). Twice daily smartphone-measurements are implemented to assess discontinuation symptoms, expectations and mood. Additionally, study visits consist of extensive measurements related to discontinuation symptoms, depressive symptomatology, psychological well-being and treatment expectations. These serve as observational measurement of different effects related to antidepressant discontinuation. During the experimental phase, outcome assessors will be blind to the randomization (i.e. treatment order) of the patients.

Objectives: At the end of the study, the investigators will determine whether open-label placebo reduces negative side effects caused by antidepressant discontinuation by aggregating the N-of-1 trials. Underlying mechanisms such as treatment expectations, as well as the relation to depressed mood, will be under explorative investigation. Additionally, the course of discontinuation symptoms, depressive symptoms (self-report and expert-rated) and treatment adherence during the entire study will be explored. Therefore, potential modulators such as psychopathology, demographics, adverse events, expectations, prior experience, subjective stress, side effects of antidepressants and anxiety vs. depression (trait/state) will be taken into account in data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18+years) with a former diagnoses of major depressive disorder (MDD), single or recurrent as main diagnosis confirmed by prescribing physician and currently remitted
* Intake of selective serotonin reuptake inhibitors (SSRI)/ serotonin-norepinephrine reuptake inhibitors (SNRI) (citalopram 20-40mg, duloxetine 60-100mg, escitalopram 10-20mg, paroxetine 20-40mg, sertraline 50-150mg, venlafaxine 75-150mg) or noradrenergic and specific serotonergic antidepressants (NaSSA) (mirtazapine 30-45mg)
* Discontinuation wish by patient supported by prescribing physician
* Fulfils the criteria of the S3 national guideline recommendations "Depression" to discontinue antidepressant medication: a) response to antidepressant; b) symptom remission for at least 4 months (first episode) or for 2 years (2 or more episodes with significant functional impairment), constant intake of antidepressant medication (at least 4 weeks on a steady dose)
* Informed consent

Exclusion Criteria:

* Current moderate or severe psychopathological symptoms or psycho-social impairments
* Acute or chronic somatic illness which might interfere with depressive disorder, antidepressant or proposed study
* Acute suicidality, psychotic symptoms, substance abuse, or addiction, current mania, or hypomania confirmed by SCID-5 or other psychopathology which might interfere with depressive disorder, antidepressant or proposed study
* Any history of bipolar disorder or psychosis confirmed by SCID-5
* Severe stressful life events (e.g., death of a family member) within six months prior to study participation
* Current pregnancy
* Insufficient German language proficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in antidepressant discontinuation symptoms assessed by the 'Generic rating scale for treatment effects' (GEEE_ACT) | Continuous measurement (2xdaily) for 8 weeks
  The generic rating scale for treatment effects item 3 assesses the current treatment effect concerning side effects (i.e. antidepressant discontinuation side-effects) on a numeric analogue scale, ranging from 0-10; higher scores indicating higher antidepressant discontinuation symptoms.

SECONDARY OUTCOMES:
Change in treatment expectations assessed by 'Generic rating scale for treatment expectations' (GEEE_EXP) | Continuous measurement (2xdaily) for 8 weeks
  The generic rating scale for treatment expectations item 3 assesses treatment expectations regarding side effects (i.e. antidepressant discontinuation side-effects) on a numeric rating scale, ranging from 0-10; higher scores indicating higher treatment expectations.
Change in (depressed) mood assessed by the 'Patient-Healthcare-Questionnaire' (PHQ-2) | Continuous measurement (2xdaily) for 8 weeks
  Self-report comprising 2 items, inquiring the degree to which an individual experiences the core symptoms of depression (i.e. anhedonia and depressed mood); items are scored on a four level Likert scale ranging from 0 (not at all) - 3 (almost constant); total score range from 0-6 (higher scores indicate a higher degree of depressed mood).

OTHER OUTCOMES:
Discontinuation symptoms - 'Discontinuation Related Signs and Symptoms Scale' (DESS) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  The discontinuation related signs and symptoms scale is a self-report questionnaire to assess discontinuation symptoms, incorporating 43 discontinuation symptoms of antidepressant with intensity ratings ranging from 0 (not present) - 3 (severe); total score range from 0-129 with higher scores indicating more severe discontinuation symptoms.
Current treatment effects - 'Generic rating scale for treatment effects' (GEEE_ACT) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  The generic rating scale for treatment effects assesses the current treatment effects (i.e. antidepressant discontinuation) regarding side effects as well as positive and negative aspects on 3 numeric rating scales with eleven response options (0-10); total score range from 0-30 with higher scores indicating higher antidepressant discontinuation effects.
Subjective depressive symptomatology - 'Beck Depression Inventory' (BDI-II) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  Self-report measure to assess depressive symptoms, including 21 items with 4 response options (0-3); total scores range from 0 - 63 (higher scores indicating higher depression severity).
Expert-rated depression severity scores - 'Montgomery-Åsberg Depression Scale' (MADRS) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  Expert-rated interview to assess the severity of depression by 10 items with up to 7 rating categories (0-6) for each item; total scores range between 0-60 with higher scores indicating more severe depression severity.
Recurrence | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  New-onset depressive episode following a period of recovery. Recurrence will be determined by BDI-II sumscore (>19) or MADRS sumscore (>21) over a period of two weeks, confirmed by SCID-5-CV section for MDD.
Mental well-being - 'Short Warwick-Edinburgh Mental Wellbeing Scale' (SWEMWBS) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  Self-report questionnaire to assess mental well-being by 7 statements about thoughts and feelings using 5 response options; total score range from 7-35 with higher sum scores reflecting a higher level of mental well-being.
Adherence - single item | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks)
  Treatment adherence assessed by a single item in the clinical interview about adherence to medication or placebo (i.e. experimental phase) intake.
Treatment expectations - 'Treatment Expectation Questionnaire' (TEX-Q) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  Self-reported measure to assess patients' treatment expectations, consisting of 15 items with 11 response options, total score range from 0-150 (higher scores implying more positive treatment expectations).
Current treatment expectations - 'Generic rating scale for treatment expectations' (GEEE_EXP) | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  The generic rating scale for treatment expectations assesses treatment expectations (i.e. antidepressant discontinuation expectations) regarding positive and negative aspects as well as side effects on 3 numeric rating scales (ranging from 0-10); total score range from 0-30 with higher scores indicating higher treatment expectations.
Pre-experiences with antidepressant discontinuation - 'Generic rating scale for previous treatment experiences' (GEEE_PRE) | Baseline
  Self-reported previous experiences with antidepressant discontinuation. If experience with antidepressant discontinuation is indicated, the following 3 items rate the experiences regarding side effects as well as positive and negative aspects on 3 numeric analogue scales (ranging from 0-10); total score range from 0-30; higher scores indicate more pre-experiences with antidepressant discontinuation effects.
Subjective Stress - 'Perceived Stress Scale' (PSS-10) | Baseline
  Self-reported measure of subjective stress, including 10 items with 5 rating categories, total scores range between 0-40; higher scores are suggestive of more subjective stress.
Anxiety vs Depression - 'State-Trait-Anxiety-Depression-Inventory' (STADI) | Baseline
  Self-report questionnaire as indicator of state and trait anxiety and depression, divided in 2 sections (state vs. trait) consisting of 20 statements with 4 response options, respectively. Total scores per scale range between 20 and 80 with higher sum scores indicating higher state/trait anxiety or depression.
Side effects of SSRIs - 'Generic Assessment of Side Effects' (GASE) | Baseline, post-antidepressant discontinuation (8 weeks after baseline)
  Self-report measure to assess side effects of antidepressant medication, including 36 items (symptom descriptions) with 4 response options. Items are additionally evaluated on their relation to antidepressant medication (Yes/ No questions). Total scores range from 0-108 (higher scores are reflective of stronger experiences of side effects).
Adverse events - single safety items | Weekly during discontinuation phase (4 weeks); biweekly during experimental phase (8 weeks); follow-up (6 months later)
  Interview-based measure assessing adverse events by 3 questions (Yes/ No questions), followed by an expert-rating of the intensity of the adverse events (1-5) and relation to treatment (1-5). Higher scores indicate more and/or a higher intensity of adverse events.
Psychopathology - 'Structured Clinical Interview for DSM-5, Clinician Version' (SCID-5-CV) | Screening
  Expert-rated semi-structured interview to assess DSM-5 diagnoses.
SSRI/SNRI blood serum level | Pre-antidepressant discontinuation (1 week after baseline); post-antidepressant discontinuation (5 weeks after baseline)
  Blood analysis assessing the blood serum level.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Tilo Kircher, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (2):
- Germany (2):
  - Philipps University Marburg Medical Center, Marburg, Hesse
  - University Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
The FAB-study is a pilotproject within a special research area funded by the DFG: TRR-SFB 289 Treatment Expectation. After deidentification, individual participant data will be shared with the TRR-SFB 289 study team and will be available for other researchers upon reasonable request. Only anonymized data in agglomerated form is used for publications. No personal data of participants will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: upon reasonable request following publication
Access Criteria: upon reasonable request following publication

REFERENCES:
- [Background] Nestoriuc Y, Pan Y, Kinitz T, Weik E, Shedden-Mora MC. Informing About the Nocebo Effect Affects Patients' Need for Information About Antidepressants-An Experimental Online Study. Front Psychiatry. 2021 Apr 27;12:587122. doi: 10.3389/fpsyt.2021.587122. eCollection 2021. PMID 33986697
- [Background] Rief, W., Nestoriuc, Y., Mueller, E. M., Hermann, C., Schmidt, K., & Bingel, U. Generic rating scale for previous treatment experiences, treatment expectations, and treatment effects (GEEE). PsychArchives. 2021 https://doi.org/10.23668/PSYCHARCHIVES.4717
- [Background] Pan Y, Meister R, Lowe B, Kaptchuk TJ, Buhling KJ, Nestoriuc Y. Open-label placebos for menopausal hot flushes: a randomized controlled trial. Sci Rep. 2020 Nov 18;10(1):20090. doi: 10.1038/s41598-020-77255-z. PMID 33208855
- [Background] Bowers HM, Kendrick T, Glowacka M, Williams S, Leydon G, May C, Dowrick C, Moncrieff J, Laine R, Nestoriuc Y, Andersson G, Geraghty AWA. Supporting antidepressant discontinuation: the development and optimisation of a digital intervention for patients in UK primary care using a theory, evidence and person-based approach. BMJ Open. 2020 Mar 8;10(3):e032312. doi: 10.1136/bmjopen-2019-032312. PMID 32152159
- [Background] Meister R, Lanio J, Fangmeier T, Harter M, Schramm E, Zobel I, Hautzinger M, Nestoriuc Y, Kriston L. Adverse events during a disorder-specific psychotherapy compared to a nonspecific psychotherapy in patients with chronic depression. J Clin Psychol. 2020 Jan;76(1):7-19. doi: 10.1002/jclp.22869. Epub 2019 Oct 1. PMID 31576565
- [Background] Shedden-Mora MC, Pan Y, Heisig SR, von Blanckenburg P, Rief W, Witzel I, Albert US, Nestoriuc Y. Optimizing Expectations About Endocrine Treatment for Breast Cancer: Results of the Randomized Controlled PSY-BREAST Trial. Clin Psychol Eur. 2020 Mar 31;2(1):e2695. doi: 10.32872/cpe.v2i1.2695. eCollection 2020 Mar. PMID 36397978
- [Background] Pan Y, Meister R, Lowe B, Winkelmann A, Kaptchuk TJ, Buhling KJ, Nestoriuc Y. Non-concealed placebo treatment for menopausal hot flushes: Study protocol of a randomized-controlled trial. Trials. 2019 Aug 16;20(1):508. doi: 10.1186/s13063-019-3575-1. PMID 31420050
- [Background] Pan Y, Kinitz T, Stapic M, Nestoriuc Y. Minimizing Drug Adverse Events by Informing About the Nocebo Effect-An Experimental Study. Front Psychiatry. 2019 Jul 25;10:504. doi: 10.3389/fpsyt.2019.00504. eCollection 2019. PMID 31427995
- [Derived] Muller A, Konigorski S, Meissner C, Fadai T, Warren CV, Falkenberg I, Kircher T, Nestoriuc Y. Study protocol: combined N-of-1 trials to assess open-label placebo treatment for antidepressant discontinuation symptoms [FAB-study]. BMC Psychiatry. 2023 Oct 13;23(1):749. doi: 10.1186/s12888-023-05184-y. PMID 37833651

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05051995/SAP_000.pdf